CLINICAL TRIAL: NCT05527249
Title: Evaluation of a Dietary Supplementation Combining Proteins and Pomegranate Extracts in Older People
Acronym: Delicens2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Delicens2021
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Healthy Aging
Keywords: safety; pomegranate extracts; protein; older people
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement group (Experimental): 20g of protein powder + 1 tablet of pomegranate extracts / day for 21 days of the dietary supplement, to be taken every day before lunch time.
  Interventions: Dietary Supplement: Dietary Supplement
- Placebo group (Placebo Comparator): 20g of protein powder + 1 tablet of maltodextrin / day for 21 days of the dietary supplement, to be taken every day before lunch time.
  Interventions: Other: Placebo of the dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — 20g of protein powder + 650mg of pomegranate extracts
  Arms: Dietary supplement group
Other: Placebo of the dietary supplement — 20g of protein powder + 650mg of maltodextrin
  Arms: Placebo group

SUMMARY:
The objective of this safety study is to evaluate the safety of a combination of proteins and pomegranate extracts in healthy subjects aged 65 years or more after 21 days of supplementation.

DETAILED DESCRIPTION:
The aim of the Delicen's project is to find an effective solution to avoid undernutrition in the elderly by proposing an assortment of food products for people who are undernourished or at risk of undernutrition. These products will be enriched with proteins and pomegranate extracts. Before to realize the impact study to test products enriched with proteins and pomegranate extracts, a safety study will be carried out.

The objective of this safety study (double-blind randomized clinical trial) is to evaluate the safety of a combination of proteins and pomegranate extracts in healthy subjects aged 65 years or more in comparing a control group consuming 20g of proteins (100% of lactoserum proteins) and 650mg of maltodextrin to a test group consuming 20g of proteins (100% of lactoserum proteins) and 650mg of pomegranate extracts after 21 days of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Woman and man, aged ≥ 65 years;
* BMI from 20 to 30 and from 21 to 30 for a person aged >70 years;
* In good general health as evidenced by medical history and physical examination;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* Fluent French speaking.

Exclusion Criteria:

* Severe psychiatric disorder or disease within 6 months before inclusion (depression, bipolar disorder, severe anxiety, psychosis, schizophrenic disorders, dementia…) or severe neurologic trouble (Alzheimer's, autism, Parkinson's disease, …);
* Cancer within less than 3 years before the screening visit (except basal cell skin cancer or squamous cell skin cancer), which in the Investigator's opinion could interfere with the results of the study;
* Subjects presenting severe gastro-intestinal, severe hepatic, severe respiratory, severe kidney or severe cardiovascular disorder or severe infection (e.g., HIV, hepatitis, …);
* Uncontrolled hormonal disorders (example: thyroid problems or Cushing's syndrome);
* Uncontrolled type 1 or 2 diabetes;
* Any clinically significant disease which in the Investigator's opinion could interfere with the safety of study participants or with the results of the study;
* Allergy or intolerance to one of the components of the administered products;
* Subjects with medications/products incompatible with the study according to the investigator (i.e: medications that could interfere with nutrient absorption);
* Subjects having participated in another clinical trial (with an investigational product) one month before the screening;
* Mental or legal incapacity, unwillingness or inability to understand or not being able to participate in the study;
* Subjects consuming ONS or protein supplements one month before the screening.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline of white blood cells (10^3/μL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of red blood cells (10^6/μL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of hemoglobin level (g/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Evolution from baseline of hematocrit level (%) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Evolution from baseline of platelet count (10^3/μL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of Uric acid (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of creatinine (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of total bilirubin (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of aspartate transaminase (U/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of alanine transaminase (U/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of total cholesterol (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of triglyceride levels (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of sodium (mmol/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of potassium (mmol/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of proteins (g/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of prealbumin (g/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of urea (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of blood sugar (mg/dL) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of alkalin phosphatase (U/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of GGT (U/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of LDH (U/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of intervention.
Change from baseline of CRP (mg/L) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of completion.
Change from baseline of weight (kg) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of completion.
Change from baseline of heart rate (bpm) at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of completion.
Change from baseline of systolic blood pressure at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of completion.
Change from baseline of diastolic blood pressure at 3 weeks | 21 days
  Comparison within and between groups after 3 weeks of completion.

SECONDARY OUTCOMES:
Number of Adverse events | 21 days
  Number of adverse events
Type of Adverse events | 21 days
  Type of adverse events
Number of Concomitant drug use | 21 days
  Number of concomitant drugs
Type of Concomitant drug use | 21 days
  Type of concomitant drugs
Compliance with therapeutic units | 21 days
  Counting of therapeutic units
Compliance with protein and/or grenade powder | 21 days
  Counting of amount of powder

CONTACTS AND LOCATIONS:
Overall Officials: Louise Deldicque, Study Director — Université Catholique de Louvain
Locations (1):
- UCLouvain - CICN, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No